CLINICAL TRIAL: NCT00577096
Title: Effects of Exercise in Combination With Epoetin Alfa During High-Dose Chemotherapy and Autologous Peripheral Blood Stem Cell Transplantation for Multiple Myeloma
Brief Title: Effects of Exercise in Combination With Epoetin Alfa
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arkansas (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Ortho Biotech Clinical Affairs, L.L.C. (Industry)
Responsible Party: Elizabeth Ann Coleman, PhD, RNP, AOCN, University of Arkansas for Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB # 29287; R01NR008937 (NIH); Ortho Biotech Clinical Affairs (Other: Ortho Biotech Clinical Affairs)
Record Dates: First submitted 2007-12-17; First posted 2007-12-19 (Estimated); Results first posted 2011-04-21 (Estimated); Last update posted 2015-04-06 (Estimated); Status verified 2015-04

CONDITIONS: Multiple Myeloma
Keywords: multiple myeloma; polysomnography; quality of life; exercise
MeSH Terms: conditions — Multiple Myeloma; Motor Activity | interventions — Epoetin Alfa; Exercise; Peripheral Blood Stem Cell Transplantation; Erythrocyte Transfusion; Thalidomide; Heparin, Low-Molecular-Weight; Platelet Transfusion; Melphalan; Vincristine; Doxorubicin; Dexamethasone; Cyclophosphamide; Etoposide; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Exercise (Experimental): Study participants were computer randomized to an individualized exercise program. Participants were stratified within Arm according to whether or not they received thalidomide with heparin, and by age (60 and younger versus older than 60)
  Interventions: Drug: Epoetin Alfa; Behavioral: Exercise; Biological: Autologous Peripheral Blood Stem Cell Transplantation; Biological: Red Blood Cell Transfusion; Drug: Thalidomide; Drug: Heparin, Low-Molecular-Weight; Biological: Platelet Transfusion; Drug: Melphalan
- usual care (Active Comparator): Study participants were asked to remain as active as possible but not prescribed an individualized exercise program. Participants were stratified within Arm according to whether or not they received thalidomide with heparin, and by age (60 and younger versus older than 60)
  Interventions: Drug: Epoetin Alfa; Drug: Total Therapy II; Biological: Red Blood Cell Transfusion; Drug: Thalidomide; Drug: Heparin, Low-Molecular-Weight; Biological: Platelet Transfusion; Drug: Melphalan

INTERVENTIONS:
Drug: Epoetin Alfa — Epoetin alfa was administered per an IRB approved algorithm to study participants when hemoglobin levels dropped during high dose chemotherapy. The usual dose is 150 units/kg og body weight, three times per week, or 40,000 units weekly, with suggested target hemoglobin range of 10-12 g/dl.
  Other Names: EPO
  Arms: Exercise
Behavioral: Exercise — A home-based individualized exercise program that incorporated aerobic and strength resistance training.
  Arms: Exercise
Biological: Autologous Peripheral Blood Stem Cell Transplantation — Standard PBSCT for multiple myeloma
  Other Names: (PBSCT)
  Arms: Exercise
Biological: Red Blood Cell Transfusion — RBC Transfusion was administered as needed
  Other Names: (RBC)
  Arms: Exercise
Drug: Thalidomide — Fifty percent of the participants received 400 mg daily
  Arms: Exercise
Drug: Heparin, Low-Molecular-Weight — Patients who received thalidomide also received prophylactic low molecular weight heparin
  Arms: Exercise
Biological: Platelet Transfusion — Platelet transfusions were administered as needed
  Arms: Exercise
Drug: Melphalan — Administered with autologous peripheralblood stem cell transplantation (PBSCT) for multiple myeloma
  Arms: Exercise
Drug: Epoetin Alfa — Epoetin alfa was administered per an IRB approved algorithm to study participants when hemoglobin levels dropped during high dose chemotherapy. The usual dose is 150 units/kg of body weight, three times per week, or 40,000 units weekly, with suggested target hemoglobin range of 10-12 g/dl
  Other Names: EPO
  Arms: usual care
Drug: Total Therapy II — Standard Induction chemotherapy care included: vincristine, doxorubicin, and dexamethasone (VAD) (0.5 mg, 10 mg/m2, and 40 mg, respectively);dexamethasone, cyclophosphamide,etoposide, and cisplatin (DCEP) (40 mg, 400 mg/m2, 40 mg/m2, and 15 mg/m2,respectively); and cyclophosphamide,doxorubicin, and dexamethasone (CAD) (750 mg/m2, 15 mg/m2, and 40 mg, respectively) for mobilization.
  Other Names: vincristine; doxorubicin; dexamethasone; cyclophosphamide; etoposide; cisplatin
  Arms: usual care
Biological: Red Blood Cell Transfusion — RBC Transfusion was administered as needed
  Other Names: RBC
  Arms: usual care
Drug: Thalidomide — Fifty percent of participants received 400 mg daily
  Arms: usual care
Drug: Heparin, Low-Molecular-Weight — Patients who received thalidomide also received prophylactic low molecular weight heparin
  Arms: usual care
Biological: Platelet Transfusion — Platelet transfusions were administered as needed
  Arms: usual care
Drug: Melphalan — Administered with autologous peripheralblood stem cell transplantation (PBSCT) for multiple myeloma
  Arms: usual care

SUMMARY:
The purpose of the study was to determine the effect of Epoetin alfa therapy (short term versus long term) with and without a home-based individualized exercise program that incorporated aerobic and strength resistance training for patients being treated with high-dose chemotherapy and autologous peripheral bloodstem cell transplantation (PBSC T) for multiple myeloma. The endpoints for the study included the number of attempts at and total number of days of stem cell collection, number of RBC and platelet transfusions during the transplantation period, time-to-recovery after transplantation, and response to intensive therapy for multiple myeloma.

ELIGIBILITY:
Inclusion Criteria:

* Those who were not at high risk for impending pathologic fracture or cord compression, as determined by magnetic resonance imaging and other radiology reports and physician assessments,and enrolled in Total Therapy treatment protocols were invited to participate in the study.

Exclusion Criteria:

Patients were excluded if they showed any of the following attributes/conditions:

* Inability to understand the intent of the study
* Current diagnosis with a major psychiatric illness
* Presence of microcytic or macrocytic anemia
* Uncontrolled hypertension
* Red cell transfusions within 2 weeks; and
* Recombinant epoetin alfa within 8 weeks of study enrollment.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2001-10; Primary Completion 2004-06 (Actual); Study Completion 2004-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sharon K Coon, Study Director — University of Oklahoma
Locations (1):
- University of Arkansas for Medical Sciences, Little Rock, Arkansas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study conducted at multiple myeloma international referral center included patients newly diagnosed & eligible for treatment with aggressive treatment. Protocol included tandem peripheral blood stem cell transplants.
Groups:
- Usual Care: Participants received standard care for multiple myeloma which included: For the Short term study: Total Therapy II Chemotherapy Regimen (See Protocol) and Stem Cell Harvest. For the Long term study: Total Therapy II Chemotherapy Regimen (See Protocol) and melphalan with autologous peripheral-blood stem cell transplantation (PBSCT). For both the short and long term studies, red blood cell (RBC) and platelet transfusions were administered as needed, in addition to Epoetic Alfa (EPO) when hemoglobin levels dropped during high dose chemotherapy. The usual EPO dose is 150 units/kg of body weight, three times per week, or 40,000 units weekly, with suggested target hemoglobin range of 10-12 g/dl. Study participants were asked to remain as active as possible but not prescribed an individualized exercise program. Participants were stratified by thalidomide administration and by age (<=60 versus >60).Participants who received thalidomide also received low-molecular weight heparin
- Exercise: Participants received standard care for multiple myeloma which included: For the Short term study: Total Therapy II Chemotherapy Regimen (See Protocol) and Stem Cell Harvest. For the Long term study: Total Therapy II Chemotherapy Regimen (See Protocol) and melphalan with autologous peripheral-blood stem cell transplantation (PBSCT). For both the short and long term studies, red blood cell (RBC) and platelet transfusions as needed, in addition to Epoetic Alfa (EPO) when hemoglobin levels dropped during high dose chemotherapy. The usual EPO dose is 150 units/kg of body weight, three times per week, or 40,000 units weekly, with suggested target hemoglobin range of 10-12 g/dl. Study participants were computer randomized to an individualized exercise program that incorporated aerobic and strength resistance training. Participants were stratified by thalidomide administration and by age (<=60 versus >60). Participants who received thalidomide also received low-molecular weight heparin.
Period: Short Term Participation
Arm/Group | Usual Care | Exercise
Started | 69 | 66
Completed | 62 | 58
Not Completed | 7 | 8
Not completed — withdrew from multiple myeloma treatment | 3 | 2
Not completed — Withdrawal by Subject | 3 | 5
Not completed — Death | 1 | 1
Period: Long Term Participation
Arm/Group | Usual Care | Exercise
Started | 34 (Only the first 34 patients who met long-term eligibility (response to EPO) were enrolled.) | 35 (Only 35 patients who met long-term eligibility (response to EPO) were enrolled.)
Completed | 34 | 35 (Sub-set of patients (n=69) who completed short term (n=120) continued in long term participation.)
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Usual Care | Exercise | Total
Number analyzed (Participants) | 69 | 66 | 135
Age, Continuous [Mean (Standard Deviation); unit: years]
  Short Term Participants | 58 (9.2) | 54.5 (10.4) | 55 (10)
  Long Term Participants | 54.4 (9.7) | 55.4 (11.4) | 55 (10.6)
Sex/Gender, Customized [Number; unit: participants]
  Male (short term study) | 13 | 12 | 25
  Female (short term study) | 22 | 19 | 41
  Male (long term study) | 24 | 23 | 47
  Female (long term study) | 10 | 12 | 22
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian (short term study) | 31 | 27 | 58
  Other (short term study) | 4 | 4 | 8
  Caucasian (long term study) | 32 | 31 | 63
  Other (long term study) | 2 | 4 | 6
Region of Enrollment [Number; unit: participants]
  United States | 69 | 66 | 135

OUTCOME MEASURES:

1. Primary Outcome: Number of Red Blood Cell Transfusions Needed to Maintain Hemoglobin Levels (Short Term)
Description: The targeted hemoglobin level for each participant was 10-12 g/dl. This is the number of red blood cell (RBC) transfusions administered to participants, as part of the investigational therapy algorithm, in an attempt to alleviate the anemia caused by multiple myeloma and high-dose chemotherapy. The numbers of RBC and platelet transfusions were obtained from the University of Arkansas for Medical Sciences blood bank.
Time Frame: up to 15 weeks
Population: For the exercise group 8 participants who entered the study were not included in the analysis (2 withdrew from myeloma treatment, 1 died, 5 withdrew from study). For the usual care group 7 were not included in the analysis (3 withdrew from myeloma treatment, 1 died, 3 withdrew from study).
Measure: Mean (Standard Deviation); unit: RBC Transfusions
Arm/Group | Usual Care | Exercise
Number analyzed (Participants) | 28 | 23
RBC Transfusions | 2.3 (2.5) | 1.8 (2.2)
Statistical Analysis 1: Comparison: Usual Care vs Exercise; The null hypothesis was that there would be no difference between groups for the number of RBC transfusions; Test type: Non-Inferiority or Equivalence — ANOVA; p < 0.025, ANOVA — Bonferroni adjusted p-value for multiple comparisons; This is minus 9 (4 exercise, 5 usual care) participants who were unresponsive to Epoetin Alfa and included participants in short and long study

2. Primary Outcome: Number of Red Blood Cell Transfusions Needed to Maintain Hemoglobin Levels (Long Term)
Description: as for outcome 1
Time Frame: up to 30 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: RBC Transfusions
Arm/Group | Usual Care | Exercise
Number analyzed (Participants) | 34 | 35
RBC Transfusions | 1.8 (2.9) | 1.0 (1.3)
Statistical Analysis 1: Comparison: Usual Care vs Exercise; The null hypothesis is that there was no difference in the number of RBC tranfusions in the exercise versus usual care groups. Data was combined from the short and long term RBC transfusions; Test type: Non-Inferiority or Equivalence — ANOVA; p < 0.025, ANOVA — Bonferroni adjusted p-value for multiple comparisons; [statistical method as in outcome 1, analysis 1]

3. Primary Outcome: Number of Platelet Transfusions Needed to Maintain Adequate Number of Platelets.(Short Term)
Time Frame: up to 15 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Platelet transfusions
Arm/Group | Usual Care | Exercise
Number analyzed (Participants) | 28 | 23
Platelet transfusions | 3.1 (3.2) | 2.3 (1.6)
Statistical Analysis 1: Comparison: Usual Care vs Exercise; Test type: Non-Inferiority or Equivalence — T-test and chi-squared test to check for equivalence of groups for age, race and gender; p < 0.025, ANOVA — Bonferroni adjusted p-value for multiple comparisons; Analysis included short and long term participants

4. Primary Outcome: Number of Platelet Transfusions Needed to Maintain Adequate Number of Platelets. (Long Term)
Time Frame: up to 30 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Platelet Transfusions
Arm/Group | Usual Care | Exercise
Number analyzed (Participants) | 34 | 35
Platelet Transfusions | 3.6 (4.5) | 2.0 (2.0)
Statistical Analysis 1: Comparison: Usual Care vs Exercise; The null hypothesis was that there would be no difference between groups for the number of platelet transfusions; Test type: Non-Inferiority or Equivalence — T-test and chi-squared to check for equivalence of groups for age, race and gender; p < 0.025, ANOVA — Bonferroni adjusted p-value for multiple comparisons; [statistical method as in outcome 1, analysis 1]

5. Primary Outcome: Number of Stem Cell Collection Attempts (Short Term)
Time Frame: up to 15 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Stem Cell Collection Attempts
Arm/Group | Usual Care | Exercise
Number analyzed (Participants) | 28 | 23
Stem Cell Collection Attempts | 1.4 (0.8) | 1.1 (0.3)
Statistical Analysis 1: Comparison: Usual Care vs Exercise; Test type: Non-Inferiority or Equivalence — ANOVA; p < 0.025, ANOVA — Bonferroni adjusted p-value for multiple comparisons; [statistical method as in outcome 1, analysis 1]

6. Primary Outcome: Number of Stem Cell Collection Attempts (Long Term)
Time Frame: up to 30 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Stem Cell Collection Attempts
Arm/Group | Usual Care | Exercise
Number analyzed (Participants) | 34 | 35
Stem Cell Collection Attempts | 1.3 (0.6) | 1.1 (0.4)
Statistical Analysis 1: Comparison: Usual Care vs Exercise; The null hypothesis was that there would be no difference between groups for the number of stem cell collection attempts; Test type: Non-Inferiority or Equivalence — ANOVA; p < 0.025, ANOVA — Bonferroni adjusted p-value for multiple comparisons; [statistical method as in outcome 1, analysis 1]

7. Primary Outcome: Total Number of Days of Stem Cell Collection (Short Term)
Time Frame: up to 15 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Usual Care | Exercise
Number analyzed (Participants) | 28 | 23
Days | 5.3 (4.0) | 4.0 (2.3)
Statistical Analysis 1: Comparison: Usual Care vs Exercise; The null hypothesis was that there would be no difference between groups for the number of days of stem cell collections; Test type: Non-Inferiority or Equivalence — T-test and chi-squared to check for equivalence of groups for age, race and gender; p < 0.025, ANOVA — Bonferroni adjusted p-value for multiple comparisons; [statistical method as in outcome 1, analysis 1]

8. Primary Outcome: Total Number of Days of Stem Cell Collection (Long Term)
Time Frame: up to 30 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Usual Care | Exercise
Number analyzed (Participants) | 34 | 35
Days | 4.9 (3.1) | 4.5 (3.1)
Statistical Analysis 1: Comparison: Usual Care vs Exercise; [analysis description as in outcome 7, analysis 1]; Test type: Non-Inferiority or Equivalence — T-test and chi-squared to check for equivalence of groups for age, race and gender; p < 0.025, ANOVA — Bonferroni adjusted p-value for multiple comparisons; [statistical method as in outcome 1, analysis 1]

9. Secondary Outcome: Hemoglobin Levels Before Chemotherapy and During Transplantation Period (Short Term)
Description: Hemoglobin Levels were measured at baseline, before peripheral blood stem cell transplantation (PBSCT), During PBSCT and at hospital discharge.
Time Frame: up to 15 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: g/dl
Arm/Group | Usual Care | Exercise
Number analyzed (Participants) | 28 | 23
g/dl
  Baseline | 12.1 (1.6) | 11.6 (1.7)
  Before transplantation | 10.8 (1.5) | 11.0 (1.6)
  During transplantation | 10.1 (0.7) | 10.4 (0.9)
  At discharge | 10.6 (1.4) | 10.6 (1.1)
Statistical Analysis 1: Comparison: Usual Care vs Exercise; The null hypothesis was that there would be no difference between groups for the number of platelet transfusions; Test type: Non-Inferiority or Equivalence — T-test and chi-squared to check for equivalence of groups for age, race and gender; p < 0.025, ANOVA — Bonferroni adjusted p-value for multiple comparisons

10. Secondary Outcome: Hemoglobin Levels Before Chemotherapy and During Transplantation Period (Long Term)
Description: as for outcome 9
Time Frame: up to 30 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: g/dl
Arm/Group | Usual Care | Exercise
Number analyzed (Participants) | 34 | 35
g/dl
  Baseline | 11.5 (1.8) | 11.7 (1.8)
  Before Transplantation | 12.0 (1.6) | 12.0 (1.4)
  During Transplanation | 10.8 (1.1) | 10.8 (1.1)
  At Discharge | 10.9 (1.4) | 11.0 (1.3)

ADVERSE EVENTS:
Time Frame: up to 30 weeks
Description: All participants included in the Short and Long Term Analysis populations. Other (non-serious)Adverse Events were not collected for this study.
Arm/Group | Usual Care | Exercise
Serious Adverse Events (participants affected / at risk) | 17/62 | 25/58
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Usual Care (N=62) | Exercise (N=58)
Anemia (Blood and lymphatic system disorders) | 1 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 1
Compression fracture (Musculoskeletal and connective tissue disorders) | 0 | 1
Death (General disorders) | 1 | 1
Deep Vein Thrombosis (DVT) (Vascular disorders) | 11 | 10
Dehydration (General disorders) | 2 | 1
Fluid overload (General disorders) | 1 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 3 | 3
Hyponatremia (Blood and lymphatic system disorders) | 1 | 5
Infection / sepsis (Infections and infestations) | 5 | 1
Mucositis / diarrhea (Gastrointestinal disorders) | 1 | 1
Myocardial infarction (Cardiac disorders) | 0 | 1
Neutropenic fever (Immune system disorders) | 11 | 8
Pain (General disorders) | 1 | 1
Pneumonia (Infections and infestations) | 5 | 1
Pulmonary embolus (Vascular disorders) | 3 | 2
Rectal abcesses (Infections and infestations) | 1 | 0
Renal failure (Renal and urinary disorders) | 1 | 0
Renal stone (Renal and urinary disorders) | 1 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Ruptured diverticulum (Gastrointestinal disorders) | 0 | 1 (59)
Syncope (General disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
Patients with hemoglobin <8 g/dl received RBC transfusions according to the transplantation protocol. Analysis may have missed specific disease-related influences on hemoglobin. Randomization should have distributed disease risks equally for groups.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less